CLINICAL TRIAL: NCT01529398
Title: Efficacy of a Sensorimotor Training in Patients With Knee Osteoarthritis: a Randomized Clinical Trial
Brief Title: Sensorimotor Training Versus Resistance Training in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Aline Basolli Gomiero, Physical Therapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABG MASTER
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; exercise therapy; resistance training; proprioception
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sensorimotor training (SMT) (Active Comparator)
  Interventions: Other: Sensorimotor training (SMT)
- Resistance training (RT) (Active Comparator)
  Interventions: Other: Resistance training (RT)
- Control group (CG) (Sham Comparator)
  Interventions: Other: Control group (CG)

INTERVENTIONS:
Other: Sensorimotor training (SMT) — The group realized 16 weeks of sensorimotor training, twice a week, with duration of 30 minutes each session. The intervention included agility and coordination exercises, perturbation training and stretching exercises. Also, the participants received orientation about the knee osteoarthritis.
  Other Names: Agility/perturbation training; proprioceptive training; neuromuscular training
  Arms: sensorimotor training (SMT)
Other: Resistance training (RT) — The group realized 16 weeks of resistance training for the quadriceps and hamstring muscles, twice a week, with duration of 30 minutes each session. The intervention included strength leg raises, simple quadriceps and hamstring strengthening with cuff weights realized in 3 sets of ten repetition maximum(10RM) for each muscle group. The group also realized stretching exercises for lower limbs and received orientation about the knee osteoarthritis.
  Arms: Resistance training (RT)
Other: Control group (CG) — Patients in this group also received information about knee osteoarthritis and realized the same warm-up and cool-down intervention realized in the interventional groups. During 16 weeks they went to the ambulatory twice a week to perform 5 minutes of stationary bicycle and 5 minutes of stretching exercises for lower limbs.
  Arms: Control group (CG)

SUMMARY:
People with knee osteoarthritis (OA) have functional instability and defective neuromuscular function, it was recently suggested that sensorimotor exercises may be important and needed to improve the effectiveness of training programs for these patients. This study objective was to compare the effectiveness of a supervised resistance muscular training (RT) versus sensorimotor training (SMT) for patients with Knee OA, on decrease of pain and functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with tibiofemoral osteoarthritis;
* Both genders;
* Age> 50 years <75 years;
* Completion of clinical and radiological criteria of the American College of Rheumatology (ACR) criteria for knee OA;
* No physical activity in the previous 3 months;
* Education level from the 4th grade of primary school.

Exclusion Criteria:

* uncontrolled hypertension;
* decompensated diabetes mellitus;
* uncontrolled thyroid diseases;
* cardiorespiratory disease (ischemia, arrhythmia, chest pain, or exercise-induced bronchospasm), liver abnormalities;
* Patients with grade IV functional limitation that needed devices to walk(Kellgren-Lawrence radiographic classification);
* Patients in a period of sick leave by the INSS or any other related factor;
* Other rheumatic diseases.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale of pain (VAS) | 16 weeks
Get Up and Go Test | 16 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 16 weeks
electromyographic analysis of quadriceps muscle (EMG) | 16 weeks
isometric quadriceps strength | 16 weeks
Medical Outcomes Study Short Form (SF-36) | 16 weeks
  Generic, patient-report measure designed to assess health-related quality of life, comprises 36 items divided into 8 subscales.
  1. Physical Functioning
  2. Role Limitations due to Physical Problems
  3. General Health Perceptions
  4. Vitality
  5. Social Functioning
  6. Role Limitations due to Emotional Problems
  7. General Mental Health
  8. Health Transition
Berg Balance Test | 16 weeks
Tinetti Test | 16 weeks
activities of daily living scale (ADLS) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Virginia FM Trevisani, MD, MS, PhD, Study Director — Federal University of São Paulo and Santo Amaro University; Maria S Peccin, PT, MS, PhD, Study Chair — Federal University of São Paulo; Marcelo Abrahão, PT, Study Chair — Federal University of São Paulo; Alvaro N Atallah, MD, PhD, Study Director — Federal University of São Paulo; Aline B Gomiero, PT, Principal Investigator — Federal University of São Paulo; Andrea H Kayo, PT, MS, Study Chair — Federal University of São Paulo
Locations (1):
- Department of Rheumatology and Physiotherapy of Interlagos Ambulatory - Santo Amaro University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fitzgerald GK, Piva SR, Gil AB, Wisniewski SR, Oddis CV, Irrgang JJ. Agility and perturbation training techniques in exercise therapy for reducing pain and improving function in people with knee osteoarthritis: a randomized clinical trial. Phys Ther. 2011 Apr;91(4):452-69. doi: 10.2522/ptj.20100188. Epub 2011 Feb 17. PMID 21330451
- [Background] Fitzgerald GK, Childs JD, Ridge TM, Irrgang JJ. Agility and perturbation training for a physically active individual with knee osteoarthritis. Phys Ther. 2002 Apr;82(4):372-82. PMID 11922853
- [Background] Diracoglu D, Aydin R, Baskent A, Celik A. Effects of kinesthesia and balance exercises in knee osteoarthritis. J Clin Rheumatol. 2005 Dec;11(6):303-10. doi: 10.1097/01.rhu.0000191213.37853.3d. PMID 16371799
- [Background] Fransen M, McConnell S. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004376. doi: 10.1002/14651858.CD004376.pub2. PMID 18843657
- [Derived] Gomiero AB, Kayo A, Abraao M, Peccin MS, Grande AJ, Trevisani VF. Sensory-motor training versus resistance training among patients with knee osteoarthritis: randomized single-blind controlled trial. Sao Paulo Med J. 2018 Jan-Feb;136(1):44-50. doi: 10.1590/1516-3180.2017.0174100917. Epub 2017 Dec 7. PMID 29236934